CLINICAL TRIAL: NCT03687944
Title: The Validity and Reliability of Unsupported Upper Limb Exercise Test in Individuals With Rheumatoid Arthritis
Brief Title: Unsupported Upper Limb Exercise Test in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin,PT, PhD, Pamukkale University
Other Study IDs: 60116787-020/58593
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Unsupported Upper Limb Exercise Test; Validity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validity and reliability — Test-retest method and concurrent validity

SUMMARY:
Evaluation of upper extremity functionalities, strength and endurance of individuals with rheumatoid arthritis is important in terms of establishing treatment program and determining treatment results. In the literature, Unsupported Upper Limb Exercise Test (UULEX) has been found to be a valid and reliable method for endurance of unsupported upper extremity in individuals with chronic obstructive pulmonary disease and is frequently used to evaluate endurance in these patients. However, there is no study on the validity and reliability of UULEX in patients with rheumatoid arthritis.The aim of this study was to determine whether the Unsupported Upper Limb Exercise Test (UULEX) is a valid and reliable method to evaluate the upper extremity endurance in individual with rheumatoid arthritis (RA). To study; a minimum of 70 individual with RA under the age of 65 who are diagnosed with RA and have no other disease affecting the upper extremity performance will be included in the rheumatology outpatient clinic.The patients with upper extremity pain that will affect the performance of the upper extremity will be excluded from the study.

The tests will be done after the demographic data of the individuals are taken. Tests will be applied to individuals before application. After each test, individuals will rest for 5 minutes to reduce the effect of fatigue. The tests will take approximately 30-40 minutes to complete. For test-retest reliability, UULEX will be reapplied after one week. For compliance validity of the UULEX, Disability Assessment Shoulder and Hand Questionnaire (DASH), Health Assessment Questionnaire (HAQ), 30 sec Push up-Pull test and 6 minute pegboard and ring test will be applied.

DETAILED DESCRIPTION:
Unsupported Upper Limb Exercise Test (UULEX):Individual sit on the chair in a way that touches the wall with the lines of the UULEX. The tables of the UULEX contain 8 horizontal levels. Each level is 84 cm wide and 8 cm high. The distance between the level centers is 15 cm. The line below corresponds to the knee level of the participant. The individual moves the plastic bar, which has a weight of 0.2 kg, from the hips by holding the arms at the shoulder width and moves it to the different levels of the lines of the UULEX in front of it. Each movement starts at the hip joint and ends at the hip joint. After making the first level for two minutes, the upper levels are made in two minute. The beginning and end point of each level is the hip joint. The bar is removed until 30 movements per minute accompanied by a metronome (level up). When individuals reach their maximum height, the bar weighing 0.2 kg is replaced with a 0.5 kg weighted bar. This weight will continue to raise to the maximum height. The weight is then increased by 0.5 kg per minute to 2 kg. Individual is referred to the test to continue until symptom limitation.

Statistical Analyses:The data will be given as mean ± standard deviation (X ± SD). The Intraclass Correlation Coefficient (ICC) will be used to evaluate the reliability of the UULEX. For concurrent validity, the relationship of the 30 sec Push up-Pull Test, DASH, HAQ and the 6-peg board ring test will be evaluated with Pearson correlation analysis. In our study, 85% power was obtained in the design made with 5% type 1 error and at least 70 patients. p value will be taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis

Exclusion Criteria:

* People who are over 65 years of age, who have carpal tunnel syndrome and adherent capsule, who have undergone surgery for upper extremity, who are pregnant or can not cooperated will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Unsupported Upper Limb Exercise Test | two week
  Endurance test

SECONDARY OUTCOMES:
6 minute pegboard and ring test | one week
  endurance test

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, Dr, Study Chair — Antalya Training and Research Hospital
Locations (1):
- Pamukkale University, Denizli, Kinikli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data of individuals will be given in the spss program

REFERENCES:
- [Result] Lima VP, Velloso M, Almeida FD, Carmona B, Ribeiro-Samora GA, Janaudis-Ferreira T. Test-retest reliability of the unsupported upper-limb exercise test (UULEX) and 6-min peg board ring test (6PBRT) in healthy adult individuals. Physiother Theory Pract. 2018 Oct;34(10):806-812. doi: 10.1080/09593985.2018.1425786. Epub 2018 Jan 19. PMID 29351493